CLINICAL TRIAL: NCT01739608
Title: Assessment of the Participation Rate and the Diagnostic Accuracy of a Colorectal Cancer Screening Program: CT Colonography Versus Flexible Sigmoidoscopy. Evaluation of a New Model Based on Telediagnosis
Brief Title: Participation and Detection Rate of Screening CT Colonography and Screening Sigmoidoscopy
Acronym: Proteus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Collaborators: im3D S.p.A. (Other); Regione Piemonte (Other); Candiolo Cancer Institute - IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14334-c27.2
Record Dates: First submitted 2012-05-23; First posted 2012-12-03 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer
Keywords: CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT Colonography (CTC) (Experimental): Invitation to screening. Subject who consent to participate in the study undergo to low dose CTC examination with limited bowel preparation.
  Interventions: Other: Invitation to screening
- Sigmoidoscopy (FS) (Active Comparator): Invitation to screening. Subjects who consent to participate in the study undergo to FS.
  Interventions: Other: Invitation to screening

INTERVENTIONS:
Other: Invitation to screening — Invitation to screening

SUMMARY:
The objectives of this multicenter, randomized trial is to assess the participation rate achievable through two different screening strategies (Computed Tomographic Colonography-CTC and sigmoidoscopy-FS), to compare detection rate of colorectal cancer (CRC) and advanced adenoma of tests and to evaluate their costs. The role of Computer-aided detection (CAD) for CTC screening will be also assessed. The trial involves 10 Italian centers located in the Piedmont Region and in Verona. Residents aged 58-60 years in those districts are target for recruitment. Exclusion criteria include: previous diagnosis of cancer or adenoma; family history or hereditary syndromes; personal history of inflammatory bowel disease; patients screened by colonoscopy or FOBT within 2 years; severe disease.

DETAILED DESCRIPTION:
Design:

* To compare detection of advanced neoplasia of CT colonography (CTC) to sigmoidoscopy (FS), a total of 20.000 eligible individuals living in the target areas are mailed an invitation letter to participate in the trial. All invitees are asked to call the screening centre in order to receive detailed information about study protocol, the screening examinations and the bowel preparation. Responders who consent to participate in the study are randomly assigned to undergo screening with CTC or FS. All non-responders will be invited to Fecal Occult Blood test (FOBT) according to the current screening procedure. In the CTC arm, positive patients (containing at least one polyp 6 mm or larger) are referred to colonoscopy; negative patients (no polyps >5 mm) are scheduled to be invited to have an FOBT after two years. In the FS arm, positive patients (at least one advanced adenoma found during FS examination) are referred to colonoscopy; negative patients are offered no further follow-up.
* To compare participation rate to FS and CTC, 1200 individuals living in the target areas and never screened for colorectal cancer, are randomly assigned to receive an invitation for screening with CTC or FS. Individuals of both groups will receive an invitation letter and an information leaflet, containing information about colorectal cancer, importance of screening, and advantages and possible risks of the selected test. Invitation letter for CTC contains a phone number of the screening centre. All invitees are asked to call the screening centre in order to receive information about bowel preparation. All non-responders will receive a remainder by mail after one month. Non-responders to reminder will be invited to FS according with current screening procedure. In the CTC arm, positive patients (containing at least one polyp 6 mm or larger) are referred to colonoscopy; negative patients (no polyps >5 mm) are scheduled to be invited to have an FOBT after two years. In the FS arm, positive patients (at least one advanced adenoma found during FS examination) are referred to colonoscopy; negative patients are offered no further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic individuals, at average risk for CRC, 58-60 years old.

Exclusion Criteria:

* Personal history of CRC or polyps
* Family history of CRC or polyps
* A terminal illness or inflammatory bowel disease
* Previous five years complete colonoscopy or a FOBT within the previous 2 years
* Patients who are unable to give informed consent

Ages: 58 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40945 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Detection rate for cancer and advanced adenoma of CT Colonography versus FS in an invitational CRC screening program | three years
  Proportion of subjects detected with CRC or advanced adenomas out of those examined
Participation rate to FS and CT Colonography | one year
  Proportion of subjects attending the proposed examination out of those invited

SECONDARY OUTCOMES:
Number of participants with severe adverse events in both screening groups | three years
  Absolute number of events
Costs of a CRC screening based on CTC | three years
  Unit cost of each procedures for participants
Type of false positive detections of Computer-aided detection for CTC in a CRC screening program | three years
  Characteristics of false positive subjects

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Regge, MD, Principal Investigator — Institute for Cancer Research and Treatment at Candiolo
Locations (1):
- S.C.D.O. Epidemiologia dei Tumori - Azienda Ospedaliera S. Giovanni Battista di Torino, Turin, Piedmont, Italy

REFERENCES:
- [Derived] Regge D, Iussich G, Segnan N, Correale L, Hassan C, Arrigoni A, Asnaghi R, Bestagini P, Bulighin G, Cassinis MC, Ederle A, Ferraris A, Galatola G, Gallo T, Gandini G, Garretti L, Martina MC, Molinar D, Montemezzi S, Morra L, Motton M, Occhipinti P, Pinali L, Soardi GA, Senore C. Comparing CT colonography and flexible sigmoidoscopy: a randomised trial within a population-based screening programme. Gut. 2017 Aug;66(8):1434-1440. doi: 10.1136/gutjnl-2015-311278. Epub 2016 Apr 12. PMID 27196588
- [Derived] Regge D, Iussich G, Senore C, Correale L, Hassan C, Bert A, Montemezzi S, Segnan N. Population screening for colorectal cancer by flexible sigmoidoscopy or CT colonography: study protocol for a multicenter randomized trial. Trials. 2014 Mar 28;15:97. doi: 10.1186/1745-6215-15-97. PMID 24678896